CLINICAL TRIAL: NCT06300684
Title: Sleep, Diet and Chrononutrition: Studying the Dual Effect of Cognitive Behavioral Therapy for Insomnia (CBTi) on Sleep and Dietary Habits
Brief Title: Exploring CBTi's Dual Effect on Sleep, Diet, & Chrononutrition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBS-2022-0085
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Insomnia
Keywords: Chrononutrition; Diet; Sleep; Circadian Rhythm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This parallel-design interventional study randomly assigns participants to receive either Cognitive Behavioral Therapy for Insomnia (CBTi) or basic sleep hygiene education over four weeks. CBTi aims to enhance sleep quality, while the control group receives sleep hygiene education. Pre- and post-intervention assessments will measure sleep parameters and dietary habits, comparing outcomes between groups. Randomization ensures unbiased assignment. Statistical analysis evaluates CBTi's effectiveness in improving sleep patterns and diet, exploring the potential indirect impact of improved sleep on diet.
Who Masked: Participant
Masking Description: Participants will be blinded to the specific type of intervention they will receive, whether it is Cognitive Behavioral Therapy for Insomnia (CBTi) or basic sleep hygiene education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-i (Experimental): The CBT-i group consists of participants who will receive Cognitive Behavioral Therapy for Insomnia (CBTi) over 4 weeks (1 session per week). This intervention involves structured sessions aimed at addressing maladaptive sleep behaviors and promoting healthy sleep habits. Participants in this group will engage in cognitive restructuring, relaxation techniques, and sleep hygiene education to improve sleep quality and duration. The goal of CBTi is to modify behaviors and thoughts that contribute to insomnia, leading to more restful and consolidated sleep patterns.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-i)
- Sleep Hygiene (No Intervention): The Sleep Hygiene group consists of participants who will not receive any specific therapeutic intervention. Instead, participants in this group will receive basic sleep hygiene education, which includes general recommendations and guidance on healthy sleep habits, which does not involve a structured therapeutic intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-i) — This intervention involves structured sessions aimed at addressing maladaptive sleep behaviors and promoting healthy sleep habits. Participants in this group will engage in cognitive restructuring, relaxation techniques, and sleep hygiene education to improve sleep quality and duration. The goal of CBTi is to modify behaviors and thoughts that contribute to insomnia, leading to more restful and consolidated sleep patterns.
  Arms: CBT-i

SUMMARY:
This study aims to investigate the effects of Cognitive Behavioral Therapy for Insomnia (CBTi) on both sleep patterns and dietary habits in Lebanese adults with insomnia. Sleep patterns and dietary habits are intricately linked, with dysregulated sleep associated with poor diet quality and increased snacking. Conversely, the types of nutrients consumed can affect hormonal balance and circadian rhythm. Insomnia and obesity are interrelated public health concerns, with CBTi showing efficacy in improving sleep. This study will recruit participants with insomnia and randomly assign them to receive either CBTi or basic sleep hygiene education. Baseline assessments will include validated questionnaires about insomnia, dietary habits, and physical activity and a 7-day 24-hour diet recall sheets, as well as actigraphy for sleep parameters, and physical activity assessments. The intervention will last for four weeks, with post-intervention assessments conducted similarly to baseline.

DETAILED DESCRIPTION:
This study aims to investigate the dual effect of Cognitive Behavioral Therapy for Insomnia (CBTi) on both sleeping patterns and dietary habits in Lebanese adults with insomnia. Sleep patterns and dietary habits are known to be closely interconnected, with dysregulated sleep often associated with poor diet quality and increased snacking. Conversely, the types of nutrients consumed can influence hormonal balance and circadian rhythm, impacting overall sleep quality.

Participants meeting the criteria for insomnia will be recruited and randomly assigned to either the intervention group receiving CBTi or the control group receiving basic sleep hygiene education. Baseline assessments will include comprehensive sleep evaluations using validated measures such as the Insomnia Severity Index (ISI), Pittsburgh Sleep Quality Index (PSQI), and actigraphy for objective sleep parameters over 7 days prior to the intervention. Additionally, participants will complete 7-day 24-hour diet recall sheets to assess dietary habits. Physical activity assessments will also be conducted using the short form of the International Physical Activity Questionnaire (IPAQ). Emotional eating will also be assessed through an 18-item emotional eating questionnaire (EEQ).Patients will also complete the PHQ-4 (Patient Health Questionnaire 4) questionnaire for assessment of depression and anxiety.

During the intervention phase, participants in the treatment group will undergo Cognitive Behavioral Therapy for insomnia (CBTi) aimed at improving sleep quality, while those in the control group will receive placebo sleep intervention that consists of sleep hygiene tips. Post-intervention assessments will mirror baseline evaluations, allowing for the comparison of changes in sleep patterns and dietary habits between the two groups.

* Data collection involves the use of physical questionnaires and actigraphy devices. Paper-based data is securely stored in a locked drawer accessible only to research personnel. Actigraphy data is retrieved using specialized software, and any invalid or corrupt data prompts reassessment. Regular audits ensure data accuracy.
* Data entered into the registry undergoes thorough checks for consistency and adherence to predefined rules. Any discrepancies are flagged for further investigation and resolution.
* Validated measures such as the Insomnia Severity Index (ISI) and Pittsburgh Sleep Quality Index (PSQI) are used alongside actigraphy to ensure accurate sleep data. Multiple sources are cross-referenced to enhance data accuracy.
* Variables include diet parameters (e.g., Late-Night Eating occasions, Eating Period) and sleep parameters (e.g., Bed Time, Total Sleep Time). Each variable is clearly defined with coding information and normal ranges where applicable.
* Recruitment occurs via snowball sampling and data collection through physical questionnaires. Data is digitized and tabulated for analysis using SPSS (Statistical Package for Social Sciences). Actigraphy data is analyzed using specialized software. Adverse events are reported and managed according to established procedures.
* Sample size assessment to specify the number of participants: A total of 40 participants will be recruited for the study to ensure adequate statistical power.
* Plan for missing data: Regular audits and checks allow early identification of missing data. Participants with missing data are prompted to provide the necessary information, or alternative participants are recruited.
* Statistical analysis plan: Statistical analyses include Wilcoxon signed-rank tests to assess pre-post intervention improvements, Spearman bivariate analysis to explore correlations between diet and sleep parameters, and Mann-Whitney tests to compare intervention and control group outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English literate adult men and women participants aged 18 to 65 years with a complaint of insomnia.

Exclusion Criteria:

* Participants under 18 years old or above 65 years old.
* Participants with a known sleep disorder other than insomnia (sleep apnea, narcolepsy, or restless leg syndrome).
* Participants with a history of neurological disease including epilepsy/seizures and traumatic brain injury.
* Participants with active psychosis.
* Participants with hearing impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in Bed Time | immediately after the intervention of 4 weeks duration
  Participants undergoing Cognitive Behavioral Therapy for Insomnia (CBTi) are expected to demonstrate significant change in Bed Time (in hours).
Change in Get Up Time | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are expected to demonstrate significant improvements in Get Up Time (in hours).
Change in Time in Bed | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are expected to demonstrate significant improvements in Time in Bed (in hours).
Change in Sleep Onset Latency (in minutes). | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are expected to demonstrate significant reductions in Sleep Onset Latency (in minutes).
Change in Sleep Efficiency | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are expected to demonstrate significant improvements in Sleep Efficiency (percentage).
Change in Wake After Sleep Onset | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are expected to demonstrate significant decreases in Wake After Sleep Onset (in minutes).
Change in Late-Night Eating Occasions number | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are anticipated to demonstrate a decrease in late-night eating occasions.
Change in Eating Window Duration and Fasting Window Duration | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are anticipated to exhibit a narrower and more restricted eating window in hours and consequently an increase in the nightly fasting period.
Change in Number of Meals | immediately after the intervention of 4 weeks duration
  Participants undergoing CBTi are anticipated to experience alterations in the number of meals consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Farid Talih, MD, Principal Investigator — American University of Beirut Medical Center
Locations (2):
- Lebanon (2):
  - Lebanese American University, Byblos, Keserwan-Jbeil Governorate
  - American University of Beirut Medical Center, Beirut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuraikat FM, Wood RA, Barragan R, St-Onge MP. Sleep and Diet: Mounting Evidence of a Cyclical Relationship. Annu Rev Nutr. 2021 Oct 11;41:309-332. doi: 10.1146/annurev-nutr-120420-021719. Epub 2021 Aug 4. PMID 34348025
- [Background] Ferini-Strambi L, Auer R, Bjorvatn B, Castronovo V, Franco O, Gabutti L, Galbiati A, Hajak G, Khatami R, Kitajima T, McEvoy D, Nissen C, Perlis M, Pevernagie DA, Randerath W, Riemann D, Rizzo G, Van Someren E, Vgontzas A, Barazzoni F, Bassetti C; European Sleep Foundation. Insomnia disorder: clinical and research challenges for the 21st century. Eur J Neurol. 2021 Jul;28(7):2156-2167. doi: 10.1111/ene.14784. Epub 2021 Apr 9. PMID 33619858
- [Background] Buenaver LF, Townsend D, Ong JC. Delivering Cognitive Behavioral Therapy for Insomnia in the Real World: Considerations and Controversies. Sleep Med Clin. 2019 Jun;14(2):275-281. doi: 10.1016/j.jsmc.2019.01.008. Epub 2019 Mar 29. PMID 31029193
- [Background] Davidson JR, Dawson S, Krsmanovic A. Effectiveness of Group Cognitive Behavioral Therapy for Insomnia (CBT-I) in a Primary Care Setting. Behav Sleep Med. 2019 Mar-Apr;17(2):191-201. doi: 10.1080/15402002.2017.1318753. Epub 2017 May 2. PMID 28463015
- [Background] Siebern AT, Manber R. New developments in cognitive behavioral therapy as the first-line treatment of insomnia. Psychol Res Behav Manag. 2011;4:21-8. doi: 10.2147/PRBM.S10041. Epub 2011 Feb 25. PMID 22114532
- [Background] Duraccio KM, Zaugg K, Jensen CD. Effects of Sleep Restriction on Food-Related Inhibitory Control and Reward in Adolescents. J Pediatr Psychol. 2019 Jul 1;44(6):692-702. doi: 10.1093/jpepsy/jsz008. PMID 30861067
- [Background] Duraccio KM, Krietsch KN, Chardon ML, Van Dyk TR, Beebe DW. Poor sleep and adolescent obesity risk: a narrative review of potential mechanisms. Adolesc Health Med Ther. 2019 Sep 9;10:117-130. doi: 10.2147/AHMT.S219594. eCollection 2019. PMID 31572040
- [Background] Goldschmidt AB, Evans EW, Saletin JM, O'Sullivan K, Koren D, Engel SG, Haedt-Matt A. Naturalistic, multimethod exploratory study of sleep duration and quality as predictors of dysregulated eating in youth with overweight and obesity. Appetite. 2020 Mar 1;146:104521. doi: 10.1016/j.appet.2019.104521. Epub 2019 Nov 18. PMID 31751632
- [Background] Gupta K, Jansen EC, Campos H, Baylin A. Associations between sleep duration and Mediterranean diet score in Costa Rican adults. Appetite. 2022 Mar 1;170:105881. doi: 10.1016/j.appet.2021.105881. Epub 2021 Dec 21. PMID 34942284
- [Background] Zhao M, Tuo H, Wang S, Zhao L. The Effects of Dietary Nutrition on Sleep and Sleep Disorders. Mediators Inflamm. 2020 Jun 25;2020:3142874. doi: 10.1155/2020/3142874. eCollection 2020. PMID 32684833
- [Background] Galland L. Diet and inflammation. Nutr Clin Pract. 2010 Dec;25(6):634-40. doi: 10.1177/0884533610385703. PMID 21139128
- [Background] Ngo-Nkondjock RV, Yuntao Z, Adnan H, Adnan SM, Cheteu TMW, Li Y. The chronotype conjecture in the association between dietary carbohydrate intake and high-sensitivity C-reactive protein (hs-CRP): a cross-sectional study from NHANES 2015 data. Sleep Sci. 2021 Jan-Mar;14(1):3-10. doi: 10.5935/1984-0063.20200047. PMID 34104331
- [Background] Afaghi A, O'Connor H, Chow CM. High-glycemic-index carbohydrate meals shorten sleep onset. Am J Clin Nutr. 2007 Feb;85(2):426-30. doi: 10.1093/ajcn/85.2.426. PMID 17284739
- [Background] Du C, Almotawa J, Feldpausch CE, Folk SYL, Parag H, Tucker RM. Effects of macronutrient intake on sleep duration and quality: A systematic review. Nutr Diet. 2022 Feb;79(1):59-75. doi: 10.1111/1747-0080.12671. Epub 2021 Apr 19. PMID 33876534
- [Background] Campanini MZ, Guallar-Castillon P, Rodriguez-Artalejo F, Lopez-Garcia E. Mediterranean Diet and Changes in Sleep Duration and Indicators of Sleep Quality in Older Adults. Sleep. 2017 Mar 1;40(3). doi: 10.1093/sleep/zsw083. PMID 28364422
- [Background] Oike H, Oishi K, Kobori M. Nutrients, Clock Genes, and Chrononutrition. Curr Nutr Rep. 2014 Apr 27;3(3):204-212. doi: 10.1007/s13668-014-0082-6. eCollection 2014. PMID 25101217
- [Background] Crispim CA, Zimberg IZ, dos Reis BG, Diniz RM, Tufik S, de Mello MT. Relationship between food intake and sleep pattern in healthy individuals. J Clin Sleep Med. 2011 Dec 15;7(6):659-64. doi: 10.5664/jcsm.1476. PMID 22171206
- [Background] Nasreddine L, Naja F, Chamieh MC, Adra N, Sibai AM, Hwalla N. Trends in overweight and obesity in Lebanon: evidence from two national cross-sectional surveys (1997 and 2009). BMC Public Health. 2012 Sep 17;12:798. doi: 10.1186/1471-2458-12-798. PMID 22984791
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Kliem S, Mossle T, Klatt T, Fleischer S, Kudlacek D, Kroger C, Brahler E, Beutel ME, Wiltink J. [Psychometric Evaluation of an Arabic Version of the PHQ-4 Based on a Representative Survey of Syrian Refugees]. Psychother Psychosom Med Psychol. 2016 Sep;66(9-10):385-392. doi: 10.1055/s-0042-114775. Epub 2016 Oct 10. German. PMID 27723929
- [Background] Natale V, Plazzi G, Martoni M. Actigraphy in the assessment of insomnia: a quantitative approach. Sleep. 2009 Jun;32(6):767-71. doi: 10.1093/sleep/32.6.767. PMID 19544753
- [Background] Knutson KL, Ryden AM, Mander BA, Van Cauter E. Role of sleep duration and quality in the risk and severity of type 2 diabetes mellitus. Arch Intern Med. 2006 Sep 18;166(16):1768-74. doi: 10.1001/archinte.166.16.1768. PMID 16983057
- [Background] St-Onge MP, Grandner MA, Brown D, Conroy MB, Jean-Louis G, Coons M, Bhatt DL; American Heart Association Obesity, Behavior Change, Diabetes, and Nutrition Committees of the Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; and Stroke Council. Sleep Duration and Quality: Impact on Lifestyle Behaviors and Cardiometabolic Health: A Scientific Statement From the American Heart Association. Circulation. 2016 Nov 1;134(18):e367-e386. doi: 10.1161/CIR.0000000000000444. Epub 2016 Sep 19. PMID 27647451
- [Background] Fernandez-Mendoza J, Baker JH, Vgontzas AN, Gaines J, Liao D, Bixler EO. Insomnia symptoms with objective short sleep duration are associated with systemic inflammation in adolescents. Brain Behav Immun. 2017 Mar;61:110-116. doi: 10.1016/j.bbi.2016.12.026. Epub 2016 Dec 30. PMID 28041986
- [Background] Irwin MR, Olmstead R, Carroll JE. Sleep Disturbance, Sleep Duration, and Inflammation: A Systematic Review and Meta-Analysis of Cohort Studies and Experimental Sleep Deprivation. Biol Psychiatry. 2016 Jul 1;80(1):40-52. doi: 10.1016/j.biopsych.2015.05.014. Epub 2015 Jun 1. PMID 26140821
- [Background] Patel SR, Zhu X, Storfer-Isser A, Mehra R, Jenny NS, Tracy R, Redline S. Sleep duration and biomarkers of inflammation. Sleep. 2009 Feb;32(2):200-4. doi: 10.1093/sleep/32.2.200. PMID 19238807
- [Background] Haus EL, Smolensky MH. Shift work and cancer risk: potential mechanistic roles of circadian disruption, light at night, and sleep deprivation. Sleep Med Rev. 2013 Aug;17(4):273-84. doi: 10.1016/j.smrv.2012.08.003. Epub 2012 Nov 6. PMID 23137527
- [Background] Blask DE. Melatonin, sleep disturbance and cancer risk. Sleep Med Rev. 2009 Aug;13(4):257-64. doi: 10.1016/j.smrv.2008.07.007. Epub 2008 Dec 17. PMID 19095474
- [Background] Gildner TE, Liebert MA, Kowal P, Chatterji S, Snodgrass JJ. Associations between sleep duration, sleep quality, and cognitive test performance among older adults from six middle income countries: results from the Study on Global Ageing and Adult Health (SAGE). J Clin Sleep Med. 2014 Jun 15;10(6):613-21. doi: 10.5664/jcsm.3782. PMID 24932140
- [Background] Gillin JC. Are sleep disturbances risk factors for anxiety, depressive and addictive disorders? Acta Psychiatr Scand Suppl. 1998;393:39-43. doi: 10.1111/j.1600-0447.1998.tb05965.x. PMID 9777046
- [Background] Breslau N, Roth T, Rosenthal L, Andreski P. Sleep disturbance and psychiatric disorders: a longitudinal epidemiological study of young adults. Biol Psychiatry. 1996 Mar 15;39(6):411-8. doi: 10.1016/0006-3223(95)00188-3. PMID 8679786
- [Background] Connor J, Norton R, Ameratunga S, Robinson E, Civil I, Dunn R, Bailey J, Jackson R. Driver sleepiness and risk of serious injury to car occupants: population based case control study. BMJ. 2002 May 11;324(7346):1125. doi: 10.1136/bmj.324.7346.1125. PMID 12003884
- [Background] Kapur V, Strohl KP, Redline S, Iber C, O'Connor G, Nieto J. Underdiagnosis of sleep apnea syndrome in U.S. communities. Sleep Breath. 2002 Jun;6(2):49-54. doi: 10.1007/s11325-002-0049-5. PMID 12075479
- [Background] Rajaratnam SMW, Licamele L, Birznieks G. Delayed sleep phase disorder risk is associated with absenteeism and impaired functioning. Sleep Health. 2015 Jun;1(2):121-127. doi: 10.1016/j.sleh.2015.03.001. Epub 2015 Apr 25. PMID 29073375
- [Background] Sivertsen B, Glozier N, Harvey AG, Hysing M. Academic performance in adolescents with delayed sleep phase. Sleep Med. 2015 Sep;16(9):1084-90. doi: 10.1016/j.sleep.2015.04.011. Epub 2015 May 18. PMID 26298783
- [Background] Montie K, Quaedackers L, Perlitius V, van der Horst E, Vandenbussche N, Overeem S, Pillen S. The impact of delayed sleep phase disorder on adolescents and their family. Sleep Med. 2019 Dec;64:15-22. doi: 10.1016/j.sleep.2019.05.022. Epub 2019 Jun 22. PMID 31655320
- [Background] Reimer MA, Flemons WW. Quality of life in sleep disorders. Sleep Med Rev. 2003 Aug;7(4):335-49. doi: 10.1053/smrv.2001.0220. PMID 14505600